CLINICAL TRIAL: NCT00181688
Title: A Phase II Study of ZD1839 (Iressa) Plus Anastrozole (Arimidex) in Patients With Relapsed Ovarian Cancer
Brief Title: Iressa (ZD1839) Plus Anastrozole (Arimidex) in Patients With Ovarian Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Dana-Farber Cancer Institute (Other); Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Carolyn N. Krasner, MD, PI, Massachusetts General Hospital
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 03-250
Record Dates: First submitted 2005-09-12; First posted 2005-09-16 (Estimated); Last update posted 2012-12-05 (Estimated); Status verified 2012-12

CONDITIONS: Ovarian Cancer; Peritoneal Carcinoma; Tubal Carcinoma
Keywords: Iressa; ZD1839; Anastrozole; Arimidex
MeSH Terms: conditions — Ovarian Neoplasms | interventions — Gefitinib; Anastrozole

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Iressa (ZD1839)
Drug: Arimidex (Anastrozole)

SUMMARY:
The main purpose of this study is to determine the effects (good and bad) Iressa plus anastrozole has on patients with relapsed ovarian cancer.

DETAILED DESCRIPTION:
* Patients will receive Iressa and anastrozole orally once daily until treatment is ended. Treatment will end if any of the following occur: Unacceptable adverse effects; bowel obstruction; initiation of systemic chemotherapy; development of new ascites or pleural effusions, development of co-morbid disease or disease progression.
* Patients will be given a drug log in which to record the date and time they take their pills, as well as any symptoms and concomitant medications.
* Patients will be seen monthly for the following tests and procedures; a physical examination and repeat blood work. Patients who remain free of clinical symptoms should have repeat abdominal/pelvic CT scans and chest x-rays on an every 3 month basis.

ELIGIBILITY:
Inclusion Criteria:

* Histologic or cytologic history diagnosis of primary ovarian, primary peritoneal or tubal carcinoma
* Asymptomatic from ovarian cancer
* Evidence of recurrent ovarian, peritoneal or tubal carcinoma
* Tumor sample must be positive for ER and/or PR
* 18 years of age or older
* ECOG performance status of less than or equal to 1
* Must be able to tolerate oral intake

Exclusion Criteria:

* Known hypersensitivity to Iressa or any of the excipients of this product
* Other coexisting malignancies or malignancies diagnosed within the last 5 years
* Concomitant use of phenytoin, carbamazepine, barbiturates, rifampicin, phenobarbital or St. John's wort
* Treatment with a non-approved or investigational drug within 30 days
* Any unresolved chronic toxicity greater than CTC grad 2 from previous anticancer therapy (except alopecia)
* Incomplete healing from previous oncologic or other major surgery
* Serum creatinine level greater than CTC grade 2
* Pregnant or breast feeding
* Severe uncontrolled systemic disease
* Significant clinical disorder or laboratory finding that makes it potentially unsafe for the subject to participate
* Patients currently receiving other investigational antineoplastic agents, on systemic chemotherapy or under radiation therapy treatment
* Patients previously treated with anastrozole or other aromatase inhibitor
* Unable to tolerate oral medications
* Clinical and/or radiographic evidence of current or impending bowel obstruction

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35
Dates: Start 2003-10; Primary Completion 2006-03 (Actual); Study Completion 2006-03 (Actual)

PRIMARY OUTCOMES:
To define the median time to termination of treatment with Iressa and anastrozole in patients with asymptomatic relapsed ovarian cancer.

SECONDARY OUTCOMES:
To define the median time to progression of this patient population
to assess the tumor response and safety of this treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Carolyn Krasner, MD, Principal Investigator — Massachusetts General Hospital
Locations (2):
- United States (2):
  - Massachusetts General Hospital, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts